CLINICAL TRIAL: NCT07042425
Title: The Effect of Computer-Based Cognitive Telerehabilitation on Global Cognitive Function and Quality of Life in Elderly With Mild Cognitive Impairment
Brief Title: The Effect of Cognitive Telerehabilitation in Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IKFR.10.06.25
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Geriatrics Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Based (Experimental): An intervention group that received computer-based cognitive training with online monitoring
  Interventions: Other: Computer based cognitive telerehabilitation
- Conventional (Experimental): Control group that received conventional cognitive training by an occupational therapist
  Interventions: Other: Computer based cognitive telerehabilitation

INTERVENTIONS:
Other: Computer based cognitive telerehabilitation — An intervention group received computer-based cognitive training with online monitoring and a control group that received conventional cognitive training by an occupational therapist

SUMMARY:
A quasi-experimental single-blind controlled trial with 36 elderlies with MCI. A three times a week computer-based cognitive telerehabilitation was given to intervention group for 12 weeks. The cognitive level and quality of life state were assessed at baseline (T0), after 8 weeks (T1) and 12 weeks (T2) intervention time points, using the Montreal Cognitive Assessment Indonesian version (MoCA-INA) and EuroQoL 5 Dimensions (EQ-5D) consecutively.

DETAILED DESCRIPTION:
This study aims to determine the effect of computer-based cognitive telerehabilitation on cognitive function and quality of life of elderly with mild cognitive impairment (MCI). Subjects were divided into two groups: an intervention group that received computer-based cognitive training with online monitoring and a control group that received conventional cognitive training by an occupational therapist. The examination included assessment of sarcopenia, frailty, cognitive function with MoCA-INA, and quality of life with EQ5D. The training was carried out three times per week for 12 weeks. Evaluation was carried out after week 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

• MCI with MoCA-INA score between 18 - 25, independent in doing activities of daily living.

Exclusion Criteria:

• Elderly with pre-existing neurological disorders such as stroke, Parkinson's disease, traumatic brain injury, significant clinical mental issues, major visual and/or auditory impairments, or a history of substance abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function Elderly with Mild Cognitive Impairment | 12 weeks
  Cognitive Function assessed using Montreal Cognitive Assessment Indonesian Version (MoCA-INA) - score in numerical 0-30
Quality of Life Elderly with Mild Cognitive Impairment | 12 weeks
  Quality of Life assessed using EuroQol 5 Dimensions (EQ-5D) - score in numerical 0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Sadikin Hospital, Bandung, Indonesia

IPD SHARING:
Plan to Share IPD: No